CLINICAL TRIAL: NCT05469529
Title: Comparison of Effects of Intrathecal Hyperbaric Bupivacaine Alone Versus Hyperbaric Bupivacaine Combined With Dexmedetomidine in Cesarean Section Deliveries
Brief Title: Bupivacaine Alone vs Bupivacaine and Dexmed in Cesarean Deliveries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KRL Hospital, Islamabad (Other)
Responsible Party: Principal Investigator, Rida Amjad Qureshi, Resident Anaesthesia, KRL Hospital, Islamabad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Dexmed 1
Record Dates: First submitted 2022-06-30; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine (No Intervention): Participants to be given 2ml of 0.5% bupivacaine intrathecally for elective cesarean section deliveries.
- Bupivacaine + Dexmedetomidine (Active Comparator): Participants to be given 5mcg dexmedetomidine in addition to 2ml of 0.5% bupivacaine intrathecally for elective cesarean section deliveries.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — 5mcg dexmedetomidine to be given intrathecally along with 0.5% bupivacaine.
  Other Names: Precedex
  Arms: Bupivacaine + Dexmedetomidine

SUMMARY:
The purpose of the study is to compare the onset and duration of sensory and motor block after spinal anesthesia between intrathecal bupivacaine alone vs intrathecal bupivacaine and dexmedetomidine combination.

DETAILED DESCRIPTION:
After approval from hospital ethical committee, parturient scheduled for elective Cesarean delivery falling in ASA II status, aged 18 - 45, with a BMI of 18-35kg/m2 will be allocated to either of the two groups B and D according to systemic randomized sampling technique, with every 3rd patient being enrolled in the study. The patients falling on odd numbers will be allocated group B and those falling on even numbers will be allocated group D. Written informed consent will be taken for enrollment in study. Performa questionnaire data will be collected by researcher herself (Annexure VII).

All parturients will be premedicated with Tab Omeprazole 20mg at 6:00 hours with a sip of water. Two 18G IV cannulas will be maintained in Operation Theater (OT). All patients will be pre-hydrated with Lactated Ringer's solution at rate of 20ml/kg by OT staff. On arrival to operating room standard monitoring consisting of pulse-oximeter, non-invasive blood pressure (NIBP) and ECG will be attached and baseline readings checked and recorded.

Intrathecal drugs will be prepared by the researcher herself. Patient's back will be prepared using aseptic measures, L3-L4 space will be identified and local anesthetic infiltrated. After 2 min 25 gauge pencil point spinal needle of B-Braun will be introduced. After obtaining free flow of CSF 2ml of 0.5% hyperbaric Bupivacaine 2 ml will be injected to Group B and 2ml of 0.5% bupivacaine mixed with 5µg dexmedetomidine will be injected in Group D, patient will be immediately placed in supine position. Timer will be started by the OT assistant as soon as the drug is injected. Spinal puncture will be performed by Trainee researcher herself who had experience of more than 200 spinal blocks.

Data collection will be done by fellow colleague of equal experience. Sensory blockade will be tested using pinprick method with a blunt 27G hypodermic needle every 1 min till loss of sensation at xiphoid (T6 level). Quality of motor blockade will be assessed by modified Bromage scale (Annexure I) at 3 mins then every 1 min till Bromage I motor block is achieved. Intra-operative hypotension (decrease in mean BP of more than 20%) will be treated with 3 - 6 mg ephedrine and bradycardia (HR < 60bpm) will be treated with 0.4mg atropine. Post-operative analgesia will be assessed half hourly for the 1st 3 hours, then 1 hourly using visual analogue scale (0-10) till the time to 1st request for analgesics or VAS ≥ 4, whichever comes first. Injection tramadol 50mg and injection paracetamol 1g will be used as rescue analgesia. Injection paracetamol will be given 6 hourly after the first dose for 24 hours. Duration of motor block will also be assessed via the Bromage Score along with assessment of VAS score. Time to regaining of the full flexion of knees and hips will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant females of age 18-45 years
2. ASA physical status II
3. Body Mass Index (BMI) of 18-35 kg/m2

Exclusion Criteria:

1. Any relative or absolute contra-indication to spinal anesthesia
2. Allergy to dexmedetomidine
3. Subjects with pre-existing non-obstetric medical co-morbidities
4. Patient refusal for spinal technique
5. Obstetrics emergencies

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-09-15 (Estimated); Study Completion 2022-10-15 (Estimated)

PRIMARY OUTCOMES:
Onset of Sensory Block | 8 mins
  Mean time to loss of sensation to pin prick using a 27 G blunt needle at the level of the xiphoid (T6) from the time of injection of drug intrathecally.
Onset of Motor Block | 8 mins
  Mean time taken to reach Bromage Score I from the time of injection of drug intrathecally
Duration of Sensory Block | 8 hours
  Mean time from spinal injection to the 1st request for analgesics or VAS ≥ 4; whichever comes first.
Duration of Motor Block | 8 hours
  Mean time from spinal injection to regaining of Bromage score 4

CONTACTS AND LOCATIONS:
Overall Officials: Rida Qureshi, Principal Investigator — KRL Hospital, Islamabad
Locations (1):
- KRL Hospital, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No